CLINICAL TRIAL: NCT05009420
Title: Validation of Avocatin b as a Biomarker of Food Intake for Assessing the Acute Consumption of Avocado in Free-living Individuals
Brief Title: Validation of Avocatin b as a Biomarker of Food Intake
Acronym: AVOC5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-2021-108
Record Dates: First submitted 2021-08-02; First posted 2021-08-17 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: avocado

STUDY DESIGN:
Intervention Model Description: Identify avocatin b (C17 lipid) in plasma of individuals that consumed 1 avocado
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avocado (Experimental): Identify avocatin b (C17 lipid) in plasma of individuals that consumed 1 avocado.
  Interventions: Other: Avocado

INTERVENTIONS:
Other: Avocado — avocado served with crackers as breakfast

SUMMARY:
The primary objectives are to

* Identify avocatin b (C17 lipid) in plasma of individuals that consumed 1 avocado.
* Confirm no avocation b present in the plasma of individuals that avoided avocado intake for 7 days.
* Determine the effect of an overnight fast on avocation b detection.

DETAILED DESCRIPTION:
The proposed study will be conducted in humans according to Good Clinical Practice (GCP) guidelines. All subjects will review and sign an Informed Consent Form approved by the Illinois Institute of Technology's Institutional Review Boards (IRB) prior to screening. SCREENING To learn more about the study and to pre-qualify, potential subjects can call the CNRC or visit the website posted on recruitment flyers or from other recruitment materials. If they call the CNRC, a staff member will provide a brief background on the study and ask a series of questions from a screening questionnaire to see if they may be eligible to participate. The same questionnaire is available on the website and can be filled out by potential subjects online. The screening questionnaire includes self-reported information about health status and lifestyle factors that can be used to determine if someone is not eligible for the study (i.e.: has diabetes, cardiovascular disease, on interfering meds, etc…).

Based on the results of the questionnaires, BMI calculation, and health evaluation, subjects who meet the inclusion and exclusion criteria will be invited to participate in the study. Eligible subjects will be trained on "how to prepare for study visit". This will include instructions for avoiding avocados for at least 7 days prior to the study Visit, fasting overnight (10-12 hours), avoidance of vigorous physical activity, alcoholic and caffeinated beverage consumption for at least 24 hours preceding a study day, maintain regular sleep pattern. If the subject did not get enough sleep during the night preceding a study day, the investigators will reschedule their study day.

STUDY DAY:

Study Day visit will last about 1.5 hours with a 30 minutes follow-up visit 24 h after the start of the study treatment.

On a Study Day visit, subjects will arrive at the clinic after fasting for at least 10 hours and in a well-hydrated and well-rested state. Subjects will be inquired for compliance to avocado-free food at least 7 days prior to study day and details of food intake in the 24-hour period prior to the visit to ensure consistency and compliance with the protocol requirements. After confirming compliance with the [ protocol, anthropometric measurements, vital signs (blood pressure, heart rate, and ear temperature) will be taken.

A finger prick for fasting blood glucose will be done to confirm the fasting status. A licensed healthcare professional (LHCP) will draw a baseline blood sample using a butterfly needle (Timepoint t=0). After completing a baseline blood draw, subjects will receive an avocado and crackers to eat onsite. After consuming the avocado and crackers, subjects will be given a take-home snack and be discharged and scheduled to come to CNR the following day for an additional blood sample. The subject will be instructed to fast overnight (10-12 hours), and the blood collection time will be anchored to 24 h after the start of the study treatment (avocado).

Blood collection: Blood will be collected a total of 2 times during the entire study period. The investigators will collect 4 mL of blood each time. Over the course of the whole study, the total amount of blood collected will be 8 mL, which is way less than what is allowed for a one-time blood donation (~550 mL).

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-35
* Males/females
* 25-70 years of age

Exclusion Criteria:

* Does not eat avocados for a reason prohibiting them from being willing to eat 1 avocado
* Sensitive/allergic to avocados
* Allergies to latex or oral allergy syndrome
* Unstable medical conditions such as on dialysis for renal disease, cardiac, gastrointestinal, or hepatic disease, cancer (non-melanoma skin cancer >5 years ago acceptable, any cancer site >10yrs without recurrence).
* Pregnant, lactating, intention of pregnancy
* Lost or gained 15 lbs of body weight in last 2 months
* Following restricted or weight loss dietary patterns
* Elevated alcohol intake (7+ drinks/week females; 14+ drinks/week males)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
changes in avocatin b (C17 lipid) concentration in plasma in healthy individuals, 24 hours after consumed 1 avocado. | baseline (time point 0) to 24 hours
  fasting blood sample before eating a avocado compare with fasting blood sample 24 hours after consumed 1 avocado.

SECONDARY OUTCOMES:
avocatin b (C17 lipid) concentration in plasma of individuals that avoided avocado intake for 7 days | Day-7-Day0
  fasting blood sample after avoiding avocado for 7 days from healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No